CLINICAL TRIAL: NCT06431919
Title: Carvedilol + Simvastatin vs. Carvedilol Alone for Chronic Liver Disease and Cirrhotic Cardiomyopathy and Its Impact on Hepatic Decompensation and Survival; a Double-blind Randomized Controlled Trial
Brief Title: Carvedilol + Simvastatin vs. Carvedilol Alone for Cirrhosis and Cirrhotic Cardiomyopathy and Impact on Hepatic Decompensation and Survival
Acronym: CIRROSTAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Madhumita Premkumar, ADDITIONAL PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/HEP/000214; IIRPSG-2024-01-02107 (Other Grant/Funding Number: Indian Council of Medical Research)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Decompensated Cirrhosis; Cirrhotic Cardiomyopathy; Cirrhosis, Liver; Left Ventricular Diastolic Dysfunction; Acute Kidney Injury
Keywords: Decompensated Cirrhosis; Cirrhotic Cardiomyopathy; Left ventricular diastolic dysfunction; Acute kidney injury
MeSH Terms: conditions — Liver Cirrhosis; Ventricular Dysfunction, Left; Acute Kidney Injury | interventions — Simvastatin; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Simvastatin + Carvedilol-arm (Experimental): * Simvastatin fixed dose of 20 mg per day
  * Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate
  * Standard Medical Therapy
  Interventions: Drug: Simvastatin 20mg; Drug: Carvedilol 3.125 mg
- Active Comparator: Carvedilol arm (Active Comparator): * Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate
  * Standard Medical Therapy
  Interventions: Drug: Carvedilol 3.125 mg

INTERVENTIONS:
Drug: Simvastatin 20mg — Simvastatin fixed dose of 20 mg per day
  Arms: Experimental: Simvastatin + Carvedilol-arm
Drug: Carvedilol 3.125 mg — Carvedilol: Starting dose of 3.125 mg twice daily targeted upwards q 7 days to achieve target heart rate

SUMMARY:
Cirrhosis and portal hypertension are associated with a hyperdynamic circulation and decompensation events, including development of ascites, variceal bleeding, acute kidney injury, and susceptibility to infections.

Rationale:

Cirrhosis and portal hypertension are associated with a hyperdynamic circulation and decompensation events, including ascites, variceal bleeding, acute kidney injury, and susceptibility to infections. CCM, present in 30-70% of patients, is characterized by structural and functional abnormalities in the heart, and is associated with progression of cirrhosis, impaired quality of life and poor survival. Statins play a crucial role in reducing proatherogenic LDL cholesterol levels, making them a cornerstone in managing diabetes and cardiovascular diseases (CVDs) with the aim of decreasing or reversing atherosclerosis. This trial aims to evaluate the impact and safety of simvastatin in cirrhotic cardiomyopathy.

Novelty: Simvastatin might be of special value in diastolic dysfunction through its hemodynamic and functional effects on LV remodeling and improve portal hemodynamics through the pleotropic effects of lipophilic statins.

Objectives:

The primary objective is to assess the combined effects of carvedilol and simvastatin in managing CCM vs carvedilol alone for a composite outcome to prevent decompensation and reduce all-cause mortality. We will comprehensively evaluate cardiac function, decompensation events and survival based on impact of simvastatin over the standard betablocker carvedilol.

Methods:

This is a double-blinded randomized placebo-controlled trial involving patients diagnosed with CCM. Clinical data, including cardiac imaging, cardiac biomarkers, and survival outcomes, will be assessed for either group.

Expected Outcome:

The investigators anticipate that the synergistic use of simvastatin and carvedilol will effectively reduce portal pressure, improve portal haemodynamic, and enhance cardiac remodelling. Successful reversal of LVDD can potentially prevent clinical events such as ascites, encephalopathy, and acute kidney injury (AKI).

DETAILED DESCRIPTION:
Cirrhotic cardiomyopathy (CCM) in chronic liver disease is seen as a blunted contractile responsiveness to stress, and/or altered diastolic relaxation with electrophysiological abnormalities, in absence of known cardiac disease. Cirrhosis induces systemic inflammation, and oxidative stress leading to cardiac structural remodeling, including fibrosis, hypertrophy, and chamber dilation. CCM is associated with risk of LVDD which further lead to hepatorenal syndrome (HRS), septic shock. and peri transplant cardiac complications. Autonomic dysfunction, and neurohormonal imbalances, cardiac arrhythmias, overt heart failure are common features of CCM in advanced liver disease. Efforts to ameliorate the abnormalities associated with CCM are crucial and necessitate a significant evidence-based therapeutic intervention. We have tested the use of carvedilol in this population and found that it causes an improvement in survival.

CCM can be managed by reducing preload (though nitrates), and by ameliorating neurohormonal activation. Lowering the heart rate to 55-65 beats per minute (bpm), as done with β-blockers, is likely to help by improving myocardial oxygen demand and coronary perfusion time with independent effects on portal hypertension, and heart failure. β-blockers may reduce myocardial contractility and patients with cirrhosis have low tolerance to β-blocker dosages required to achieve a THR of 55-65 bpm. Ivabradine is useful in a subset with baseline tachycardia but does not offer survival benefit over carvedilol alone. Therefore, there is a great need to evaluate other agents that can achieve improvement in CCM related complications in cirrhosis.

* Furthermore, β-blockers might diminish myocardial contractility, and patients with cirrhosis may struggle to tolerate β-blocker doses necessary for attaining a target heart rate (THR) of 55-65 bpm. Hence, there's a critical necessity to assess alternative agents capable of ameliorating complications associated with cirrhotic cardiomyopathy (CCM).
* Early interventions to avert cardiovascular morbidity will prove to be cost effective in managing outcome, as they avert high cost of managing the public health burden of all-cause mortality in cirrhosis.
* Cardiovascular complications stand as the primary cause of mortality post-liver transplantation (LT), underscoring the need for thorough evaluation before LT.
* This study will systematically screen participants for coronary artery disease as an integral part of its screening process.
* Statins, particularly simvastatin, exert a favorable impact on vascular reactivity especially in cirrhosis. Simvastatin increases the production of nitric oxide(NO), leading to increased hepatic blood flow and reduced sinusoidal resistance, particularly upon short-term exposure. resistance.
* Simvastatin has an acceptable adverse event profile in decompensated Child B patients. There is no high-quality evidence specifically evaluating the role of simvastatin in cirrhotic cardiomyopathy, although there are data to suggest its efficacy in portal hypertension. The proposed project covers an area of overlap between cardiovascular and liver disease outcomes, which reflect as decompensation events, worsening in liver severity scores and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-65 years
* Compensated cirrhosis, as diagnosed by histology or clinical, laboratory and USG findings,
* CCM (with EF>50%) on 2D echocardiography with TDI
* Written informed consent.

Exclusion Criteria:

* Age >65 years
* Serum Creatinine>2 mg/dl
* Patient previously treated with statin (one month before the study)
* Contraindications to statins
* Advanced Cirrhosis (CTP score>9)
* Coronary artery disease
* Sick sinus syndrome/ Pacemaker, valvular heart disease
* Cardiac rhythm disorder, Peripartum cardiomyopathy
* Portopulmonary hypertension/ hepatopulmonary syndrome
* Transjugular intrahepatic portosystemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Pregnancy or lactation
* Patients with HIV or retroviral therapy
* Anemia Hb < 8gm/dl in females, and < 9 gm/dl in males
* Acute variceal bleeding in last 6 months.
* Need for medications, metabolized by CYP3A4(such as amlodipine, verapamil, fenofibrate azole antibiotics, protease inhibitors etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Time to acute decompensation event | 1 Year
  The primary outcome measure is defined as a composite end point of acute decompensation event (acute variceal bleeding, new ascites or recurrence of previously controlled ascites, episode of hepatic encephalopathy or acute kidney injury) OR all-cause death in patients with cirrhosis and cirrhotic cardiomyopathy

SECONDARY OUTCOMES:
All-cause Mortality | From enrollment until 1 year of follow up
Any New decompensation event | 1 Year
  New decompensation events are defined as decompensation event( ascites, hepatic encephalopathy, variceal bleeding) in a previously compensated patient with cirrhosis or further decompensation when a new event [recurrence of ascites, hepatorenal syndrome-acute kidney injury (HRS-AKI), hepatic encephalopathy (HE), or acute variceal bleeding (AVB), spontaneous bacterial peritonitis (SBP)] occurs in a patient with previously decompensated disease
Improvement in CCM parameters (left ventricular diastolic function) in either arm based on Echocardiography and Cardiac Imaging | 1 Year
Episodes warranting hospitalization | 1 Year
  Number of hospital admissions on follow up.
Serum level of BNP and other cardiac and inflammatory biomarkers | 1 Year
  ELISA or autoanalyzer will be performed for qunatification

CONTACTS AND LOCATIONS:
Overall Officials: Dr Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Department of Hepatology, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No